CLINICAL TRIAL: NCT00514280
Title: Tobacco Smoke and Lead Exposure During Pregnancy: Intervention to Reduce Effects on Birth-Weight and Gestational Age
Brief Title: Tobacco Smoke and Lead Exposure During Pregnancy
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907199; 07-CH-N199
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-11

CONDITIONS: Lead Exposure in Pregnant Women; Tobacco Smoke Exposure Pregnant Women
Keywords: Lead and Smoke Study in D.C.; Birth Weight; Gestational Age; Lead; Tobacco Smoke
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will test whether a short interview session about lead and secondhand tobacco smoke can help pregnant women reduce their exposure to lead and secondhand smoke. Both lead and secondhand tobacco smoke can cause problems with a pregnancy. The best way to prevent exposure to lead and secondhand tobacco smoke is to recognize the sources and avoid them.

Non-smoking African-American and Hispanic pregnant women between 18 and 49 years of age who live in Washington, D.C. may be eligible for this study.

Participants are randomly assigned to one of two study groups. Both groups have a 30-minute one-on-one session with a member of the study staff. The content of the session differs between groups. In addition, all women undergo the following tests and procedures:

* Answer questions about themselves, their pregnancies, diet, home and smokers in the home.
* Requested to provide permission to obtain medical records of children older than 12 months of age who have ever been seen at Children's National Medical Center.
* Blood draws at least four times during the study: at the time of enrollment, during the second trimester of the pregnancy, during the third trimester, and at the time of delivery. Up to three optional blood samples may also be requested, one during each trimester of the pregnancy. Blood samples are used to measure lead, cotinine (a chemical the body makes out of nicotine) and hematocrit (a test for anemia).
* Collection of umbilical cord blood at the time of delivery.
* Answer questions after the delivery about the patient's health, the delivery and the baby.

DETAILED DESCRIPTION:
Prenatal exposure to lead and tobacco has been shown to cause long-term adverse effects to the fetus and child, including decreased birthweight and premature delivery. These effects have been shown even at very low exposure levels. Since both exposures can be modified, many experts recommend screening for and counseling to prevent or reduce these exposures as part of routine prenatal care. The high infant mortality in the District of Columbia (DC) (10.2 deaths per 1,000 live births, versus 6.2 deaths per 1,000 births nationally) is incompletely understood, but disparities in health and healthcare access for minority populations, premature delivery, and low birthweight are likely contributors. Several studies and prevention programs have addressed smoking by and secondhand tobacco smoke (SHS) exposure of pregnant women living in DC in an effort to reduce the infant mortality rate, but none have addressed elevated blood lead levels (BLL) or the effects of exposure to both elevated BLL and SHS. Since DC children have high rates of both elevated BLL and SHS exposure, compared to the US population, we hypothesize that pregnant women in DC have similar high rates of elevated BLL and SHS exposure, AND that these exposures contribute to the high rates of low birthweight and decreased gestational age, and therefore to the rate of infant mortality in DC. The primary aim of this study is to determine the effectiveness of a screening and secondary prevention intervention for elevated blood lead and SHS exposure of low income, pregnant women living in Washington, DC.

ELIGIBILITY:
* INCLUSION CRITERIA:

Female

Pregnant

Age 18-49

Self-identified as African-American or Hispanic/Latino

Patient at participating clinic

DC resident at the time of enrollment

No tobacco use of any kind after week 13 of the current pregnancy

Able to read, write and understand English

Able to give informed consent

Able to cooperate with testing procedures

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-08-02; Study Completion 2011-05-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States

REFERENCES:
- [Background] Haddow JE, Knight GJ, Palomaki GE, McCarthy JE. Second-trimester serum cotinine levels in nonsmokers in relation to birth weight. Am J Obstet Gynecol. 1988 Aug;159(2):481-4. doi: 10.1016/s0002-9378(88)80114-5. PMID 3407708
- [Background] Gonzalez-Cossio T, Peterson KE, Sanin LH, Fishbein E, Palazuelos E, Aro A, Hernandez-Avila M, Hu H. Decrease in birth weight in relation to maternal bone-lead burden. Pediatrics. 1997 Nov;100(5):856-62. doi: 10.1542/peds.100.5.856. PMID 9346987
- [Background] Mannino DM, Homa DM, Matte T, Hernandez-Avila M. Active and passive smoking and blood lead levels in U.S. adults: data from the Third National Health and Nutrition Examination Survey. Nicotine Tob Res. 2005 Aug;7(4):557-64. doi: 10.1080/14622200500185264. PMID 16085527